CLINICAL TRIAL: NCT00323960
Title: Five-year Single-blind, Phase III Effectiveness Randomised Actively Controlled Clinical Trial in New Onset Juvenile Dermatomyositis: Prednisone Versus Prednisone Plus Cyclosporine a Versus Prednisone Plus Methotrexate
Brief Title: Five-year Actively Controlled Clinical Trial in New Onset Juvenile Dermatomyositis
Acronym: PRINTOJDMTR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Pediatric Rheumatology International Trials Organization (Other)
Responsible Party: Principal Investigator, Nicolino Ruperto, MD, MPH, Senior Scientist of PRINTO, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGG-PRINTO-002; AIFA (Other Grant/Funding Number: Agenzia Italiana del Farmaco (no FARMJWPZ)); Myositis Association (Other Grant/Funding Number: Myositis Association)
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Juvenile Dermatomyositis
Keywords: Juvenile dermatomyositis; randomised actively controlled clinical trial; prednisone; cyclosporine; methotrexate; effectiveness
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylprednisolone pulse (MPDN)+PDN+CSA (Active Comparator): MPDN= methylprednisolone pulse PDN= prednisone or equivalent CSA= cyclosporine A
  Interventions: Drug: 3 MPDN pulse + PDN + CSA
- MPDN+PDN+MTX (Active Comparator): MPDN= methylprednisolone pulse PDN= prednisone or equivalent MTX= methotrexate
  Interventions: Drug: 3 MPDN pulse + PDN + MTX
- MPDN+PDN (Active Comparator): MPDN= methylprednisolone PDN= prednisone or equivalent
  Interventions: Drug: 3 MPDN pulse + PDN

INTERVENTIONS:
Drug: 3 MPDN pulse + PDN — 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years.
  Arms: MPDN+PDN
Drug: 3 MPDN pulse + PDN + CSA — 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Cyclosporine 5 mg/Kg/day in 2 oral doses
  Arms: Methylprednisolone pulse (MPDN)+PDN+CSA
Drug: 3 MPDN pulse + PDN + MTX — 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Methotrexate 15-20 mg/m2 once per week. Patients treated with MTX will receive concomitant folic or folinic acid according to the attending physician decision.
  Arms: MPDN+PDN+MTX

SUMMARY:
This is a 5-year project, involving 185 partners from 46 countries ((110 in 21 European Union (EU) States and 75 in 25 extra-EU States)), with a randomised clinical trials (RCT) in juvenile dermatomyositis (JDM): 5-year phase III single-blind, RCT in children with newly diagnosed JDM: prednisone (PDN) versus PDN plus methotrexate (MTX) versus PDN plus Cyclosporine A. The trial is aimed to find out the treatment regimen associated with the lowest occurrence of flare and the lowest drug related toxicity

DETAILED DESCRIPTION:
Scientific objectives: The proposed project is aimed to improve treatment approaches for rare, severe and disabling paediatric rheumatic diseases (PRD). This goal will be achieved by the Paediatric Rheumatology International Trials Organisation (PRINTO) an international network whose main function is to provide a scientific base for current PRD treatments for which no evidence based data exist in the literature, and for drugs for which there is no support from industries.

This is a 5-year project, involving 46 countries (110 in 21 EU States and 75 in 25 extra-EU States), with a randomised clinical trials (RCT) in juvenile dermatomyositis (JDM): 5-year phase III single-blind, RCT in children with newly diagnosed JDM: prednisone (PDN) versus PDN plus methotrexate (MTX) versus PDN plus Cyclosporine A (CsA). The trial is aimed to find out the treatment regimen associated with the lowest occurrence of flare and the lowest drug related toxicity. The retention on treatment will be used as main measure of effectiveness.

Methodology: The present protocol is the natural follow up of previous work conducted by PRINTO. In particular the RCT foreseen in this protocol is modelled after the successful completion of an early phase trial with MTX in juvenile idiopathic arthritis, and will use validated JDM outcome measures for the evaluation of response to therapy.

It is the basic premise of this protocol that, without i) the involvement of the international paediatric rheumatology community, ii) the innovative type of mechanism described herein, these studies would never be conducted.

Objectives. The goals of the current protocol is therefore the natural follow-up of the objectives achieved with the previous grants and, in particular, of projects designed to discern new models for the successful conduct of clinical trials in children with rare diseases, and to develop standardized and validated measures for the evaluation of response to therapy in JDM.

The proposed trial in JDM (prednisone [PDN] versus PDN plus methotrexate [MTX] versus PDN plus cyclosporine [CsA]), should serve as a model for the successful running of early phase clinical trials for severe and disabling rare diseases of childhood.

The ultimate aim of these trials is to provide evidence-based information about the clinical utility of drugs in the management of rare paediatric conditions.

ELIGIBILITY:
Inclusion Criteria. Each patient must meet all the following criteria in order to participate in this trial:

1. Newly diagnosed and untreated children (only treatment with 1 NSAID is allowed and/or prednisone >1 mg/kg/day for no more than 1 month from diagnosis) with probable or definite diagnosis of JDM according to published (12;13). If a muscle biopsy will be performed (optional) it will be read by the pathologists of the participating centres (light and immunofluorescence). Slides of paraffin-embedded sections from all patients will be re-viewed by a blinded myopathologist at PRINTO.
2. Age at enrolment ≤ 18 years.
3. Female of child-bearing potential must have a negative pregnancy test at the beginning of the trial, and then every 3 months. If sexually active, they must agree to use adequate contraception, throughout study participation, and must have no intention of conceiving during the course of the study. Post-pubertal males must have no plans to father a child during the study and agree to use adequate birth control methods if sexually active.
4. Ability to comply with the entire study procedures, ability to communicate meaningfully with the investigational staff, competence to give written informed consent; to be applied to the parents and/or patients, as appropriate
5. Duly executed, written, informed consent obtained from the parents/patient.

Exclusion Criteria. Any of the following will exclude a patient from this trial:

1. Neutrophil count <1,500/mm3 and/or platelet count <50,000/mm3
2. Demonstration of cutaneous or gastrointestinal ulceration of JDM related pulmonary disease or cardiomyopathy at the time of diagnosis.
3. History of poor compliance.
4. Evidence of current use of alcohol or illicit drugs abuse.
5. Live vaccines not allowed during the entire duration of the trial.

Dropout Criteria. Patients will be considered "treatment failures", and dropped from the trial but included in efficacy analysis, if any of the following will occur during the active period of the trial.

1. Non compliance with study medication administration
2. Enrolment in other therapeutic trials.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2006-05-31 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2015-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolino Ruperto, MD, MPH, Principal Investigator — Istituto Giannina Gaslini _ PRINTO Senior Scientist; Alberto Martini, MD, Prof., Study Chair — Istituto Giannina Gaslini_PRINTO Chairman
Locations (1):
- Istituto Giannina Gaslini, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request to the Paediatric Rheumatology InterNational Trials Organisation (PRINTO) network as per its bylaws
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available upon request
Access Criteria: Request to the Paediatric Rheumatology International Trials Organisation (PRINTO) international coordinating centre: PRINTO@gaslini.org
URL: https://www.PRINTO.it/

REFERENCES:
- [Background] Miller LC, Sisson BA, Tucker LB, DeNardo BA, Schaller JG. Methotrexate treatment of recalcitrant childhood dermatomyositis. Arthritis Rheum. 1992 Oct;35(10):1143-9. doi: 10.1002/art.1780351006. PMID 1418005
- [Background] Al-Mayouf S, Al-Mazyed A, Bahabri S. Efficacy of early treatment of severe juvenile dermatomyositis with intravenous methylprednisolone and methotrexate. Clin Rheumatol. 2000;19(2):138-41. doi: 10.1007/s100670050032. PMID 10791626
- [Background] Heckmatt J, Hasson N, Saunders C, Thompson N, Peters AM, Cambridge G, Rose M, Hyde SA, Dubowitz V. Cyclosporin in juvenile dermatomyositis. Lancet. 1989 May 13;1(8646):1063-6. doi: 10.1016/s0140-6736(89)92456-2. PMID 2566009
- [Background] Pistoia V, Buoncompagni A, Scribanis R, Fasce L, Alpigiani G, Cordone G, Ferrarini M, Borrone C, Cottafava F. Cyclosporin A in the treatment of juvenile chronic arthritis and childhood polymyositis-dermatomyositis. Results of a preliminary study. Clin Exp Rheumatol. 1993 Mar-Apr;11(2):203-8. PMID 8508564
- [Derived] Ruperto N, Pistorio A, Ravelli A, Angioloni S, Martini A; Paediatric Rheumatology International Trials Organisation (PRINTO). The PRINTO juvenile dermatomyositis trial - Authors' reply. Lancet. 2016 Jun 25;387(10038):2601. doi: 10.1016/S0140-6736(16)30671-7. No abstract available. PMID 27353819
- [Derived] Dale A, Milosevic I, Goldacre B; COMPare project team. The PRINTO juvenile dermatomyositis trial. Lancet. 2016 Jun 25;387(10038):2600-2601. doi: 10.1016/S0140-6736(16)30845-5. No abstract available. PMID 27353816
- [Derived] Ruperto N, Pistorio A, Oliveira S, Zulian F, Cuttica R, Ravelli A, Fischbach M, Magnusson B, Sterba G, Avcin T, Brochard K, Corona F, Dressler F, Gerloni V, Apaz MT, Bracaglia C, Cespedes-Cruz A, Cimaz R, Couillault G, Joos R, Quartier P, Russo R, Tardieu M, Wulffraat N, Bica B, Dolezalova P, Ferriani V, Flato B, Bernard-Medina AG, Herlin T, Trachana M, Meini A, Allain-Launay E, Pilkington C, Vargova V, Wouters C, Angioloni S, Martini A; Paediatric Rheumatology International Trials Organisation (PRINTO). Prednisone versus prednisone plus ciclosporin versus prednisone plus methotrexate in new-onset juvenile dermatomyositis: a randomised trial. Lancet. 2016 Feb 13;387(10019):671-678. doi: 10.1016/S0140-6736(15)01021-1. Epub 2015 Nov 30. PMID 26645190
- See also: Web site of the international network who is conducting the trial — http://www.printo.it

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylprednisolone Pulse+Prednisone: Group 1 received 3 pulses of methylprednisolone and has been randomized to prednisone or equivalent
- Methylprednisolone Pulse+Prednisone+Cyclosporine A: Group 2 received 3 pulses of methylprednisolone and has been randomized to prednisone or equivalent plus cyclosporine A
- Methylprednisolone Pulses+Prednisone+Methotrexate: Group 3 received 3 pulses of methylprednisolone and has been randomized to prednisone or equivalent plus methotrexate
Period: Overall Study
Arm/Group | Methylprednisolone Pulse+Prednisone | Methylprednisolone Pulse+Prednisone+Cyclosporine A | Methylprednisolone Pulses+Prednisone+Methotrexate
Started | 47 | 46 | 46
Completed | 47 | 46 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MPDN+PDN: MPDN+PDN MPDN= methylprednisolone PDN= prednisone or equivalent
  3 MPDN pulse + PDN: 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years.
- MPDN+PDN+CSA: MPDN= methylprednisolone pulse PDN= prednisone or equivalent CSA= cyclosporine A
  3 MPDN pulse + PDN + CSA: 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Cyclosporine 5 mg/Kg/day in 2 oral doses
- Total: Total of all reporting groups
Arm/Group | MPDN+PDN | MPDN+PDN+CSA | MPDN+PDN+MTX | Total
Number analyzed (Participants) | 47 | 46 | 46 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 46 | 46 | 139
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — For age it is intended age at first observation
  years | 7.2 [5.1 to 10.1] | 8.9 [5.1 to 12.4] | 7.1 [4.3 to 10.4] | 7.5 [4.6 to 10.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 30 | 82
  Male | 21 | 20 | 16 | 57
Region of Enrollment [Number; unit: participants]
  Italy | 11 | 13 | 10 | 34
  Algeria | 1 | 0 | 0 | 1
  Argentina | 11 | 2 | 2 | 15
  Austria | 1 | 0 | 0 | 1
  Belgium | 3 | 0 | 3 | 6
  Brazil | 4 | 6 | 3 | 13
  Colombia | 1 | 0 | 0 | 1
  Czech Republic | 1 | 1 | 0 | 2
  Denmark | 0 | 2 | 0 | 2
  France | 3 | 10 | 11 | 24
  Germany | 2 | 0 | 1 | 3
  Greece | 0 | 1 | 1 | 2
  Israel | 0 | 0 | 1 | 1
  Latvia | 0 | 0 | 1 | 1
  Mexico | 0 | 3 | 3 | 6
  Netherlands | 1 | 1 | 2 | 4
  Norway | 2 | 0 | 0 | 2
  Serbia | 1 | 0 | 0 | 1
  Slovakia | 0 | 2 | 0 | 2
  Slovenia | 1 | 2 | 1 | 4
  Spain | 0 | 1 | 0 | 1
  Sweden | 2 | 1 | 2 | 5
  United Kingdom | 1 | 0 | 1 | 2
  United States | 0 | 0 | 1 | 1
  Venezuela | 1 | 1 | 3 | 5
disease duration [Median (Inter-Quartile Range); unit: months] | 2.6 [1.2 to 5.1] | 2.7 [1.2 to 6.2] | 2.8 [1.9 to 5.0] | 2.8 [1.3 to 5.3]

OUTCOME MEASURES:

1. Primary Outcome: Responder Status Defined as 20% Improvement in at Least 3 Core Set Variables With no More Than 1 of the Remaining Variables, (Muscle Strength Excluded), Worsened by > 30%.
Description: The PRINTO Juvenile Dermatomyositis (JDM) core set variables are:
  1. muscle strength by the mean of the Childhood Myositis Assessment Scale (CMAS);
  2. physician's global assessment of disease activity on a 10 cm Visual Analogue Scale (VAS);
  3. global disease activity assessment by the mean of the Disease Activity Index (DAS);
  4. parent's/patient's global assessment of overall well-being on a 10 cm VAS;
  5. functional ability assessment by the mean of the Childhood Health Assessment Questionnaire (CHAQ)
  6. health-related quality of life assessment.
Time Frame: 6 months
Population: Comparison between group 2 (PDN+CSA) and 3 (PDN+MTX) combined versus group 1 (PDN)
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 (MPDN+PDN): MPDN+PDN MPDN= methylprednisolone PDN= prednisone or equivalent
  3 MPDN pulse + PDN: 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years.
- Group 2 (MPDN+PDN+CSA): MPDN= methylprednisolone pulse PDN= prednisone or equivalent CSA= cyclosporine A
  3 MPDN pulse + PDN + CSA: 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Cyclosporine 5 mg/Kg/day in 2 oral doses
- Group 3 (MPDN+PDN+MTX): MPDN= methylprednisolone pulse PDN= prednisone or equivalent MTX= methotrexate
  3 MPDN pulse + PDN + MTX: 3 methylprednisolone pulses followed (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Methotrexate 15-20 mg/m2 once per week. Patients treated with MTX will receive concomitant folic or folinic acid according to the attending physician decision.
Arm/Group | Group 1 (MPDN+PDN) | Group 2 (MPDN+PDN+CSA) | Group 3 (MPDN+PDN+MTX)
Number analyzed (Participants) | 47 | 46 | 46
Participants | 24 | 32 | 33
Statistical Analysis 1: Comparison: Group 1 (MPDN+PDN) vs Group 2 (MPDN+PDN+CSA) vs Group 3 (MPDN+PDN+MTX); We calculated that a sample size of 40 patients would be needed in each study group (total 120 patients) to have 80% power for comparison of combination treatments (prednisone plus methotrexate or prednisone plus ciclosporin) with the reference treatment (prednisone alone); Test type: Superiority; p = 0.0228, Chi-squared — For multiple hypothesis testing, we used Bonferroni's correction (with n=3 posterior comparisons); To assess proportions we used the χ² test or Fisher's exact test

2. Primary Outcome: Time to Clinical Remission
Description: Clinical remission is defined as the status of inactive disease for at least 6 continuous months defined as normal muscle strength (CMAS equal to 52) and physician global assessment of disease activity equal to 0.
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: events per 1000 persons-time
Groups:
- Group 1 (MPDN+PDN): MPDN+PDN MPDN= methylprednisolone PDN= prednisone or equivalent
  3 MPDN pulse + PDN: 3 methylprednisolone pulses (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years.
- Group 2 (MPDN+PDN+CSA): MPDN= methylprednisolone pulse PDN= prednisone or equivalent CSA= cyclosporine A
  3 MPDN pulse + PDN + CSA: 3 methylprednisolone pulses (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Cyclosporine 5 mg/Kg/day in 2 oral doses
- Group 3 (MPDN+PDN+MTX): MPDN= methylprednisolone pulse PDN= prednisone or equivalent MTX= methotrexate
  3 MPDN pulse + PDN + MTX: 3 methylprednisolone pulses (30 mg/kg/pulse max 1 gram) followed by prednisone 2 mg/Kg/day to be tapered to 0.2 mg/kg/day in 6 months and then discontinued in 2 years; Methotrexate 15-20 mg/m2 once per week. Patients treated with MTX will receive concomitant folic or folinic acid according to the attending physician decision.
Arm/Group | Group 1 (MPDN+PDN) | Group 2 (MPDN+PDN+CSA) | Group 3 (MPDN+PDN+MTX)
Number analyzed (Participants) | 47 | 46 | 46
events per 1000 persons-time | 5.99 [3.00 to 11.98] | 4.95 [2.36 to 10.38] | 13.39 [8.07 to 22.21]
Statistical Analysis 1: Comparison: Group 1 (MPDN+PDN) vs Group 2 (MPDN+PDN+CSA) vs Group 3 (MPDN+PDN+MTX); We used the Kaplan-Meier method to produce survival curves (groups 1 and 2 versus group 3) and compared them with the Log-Rank test. We judged a p value less than 0·05 significant. We reported in the table the incidence rates with 95% confidence intervals of the 3 groups; Test type: Superiority; p = 0.012, Log Rank; Relative risk = 2.45, 95% CI 2-sided [1.2 to 5.0] — RR related to prednisone plus methotrexate arm (group 3) versus prednisone alone (group 1) and prednisone plus ciclosporin (group 2)

3. Secondary Outcome: Time to Major Therapeutic Changes
Description: Time to major therapeutic changes is defined as the addition of CSA or MTX or any other disease-modifying antirheumatic drug (DMARS) in any of the 3 groups or discontinuation of assigned therapy for any reason including adverse events. Retention on treatment was used as main measure of effectiveness.
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: events per 1000 persons-time
Arm/Group | Group 1 (MPDN+PDN) | Group 2 (MPDN+PDN+CSA) | Group 3 (MPDN+PDN+MTX)
Number analyzed (Participants) | 47 | 46 | 46
events per 1000 persons-time | 30.52 [21.34 to 43.65] | 17.52 [11.31 to 27.16] | 13.92 [8.65 to 22.39]
Statistical Analysis 1: Comparison: Group 1 (MPDN+PDN) vs Group 2 (MPDN+PDN+CSA) vs Group 3 (MPDN+PDN+MTX); We used the Kaplan-Meier method to produce survival curves (group 1 versus groups 2 and 3) and compared them with the Log-Rank test. We judged a p value less than 0·05 significant. We reported in the table the incidence rates with 95% confidence intervals of the 3 groups; Test type: Superiority; p = 0.009, Log Rank; Relative risk = 1.95, 95% CI 2-sided [1.2 to 3.15] — RR related to prednisone alone (group 1) versus prednisone plus ciclosporin (group 2) and prednisone plus methotrexate arm (group 3)

4. Secondary Outcome: Time to Prednisone, or Equivalent, Discontinuation
Description: Prednisone or equivalent glucocorticoid discontinuation is defined as the complete discontinuation of glucocorticoids
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: events per 1000 persons-time
Arm/Group | Group 1 (MPDN+PDN) | Group 2 (MPDN+PDN+CSA) | Group 3 (MPDN+PDN+MTX)
Number analyzed (Participants) | 47 | 46 | 46
events per 1000 persons-time | 15.91 [10.15 to 24.94] | 27.82 [19.56 to 39.55] | 24.42 [16.50 to 36.14]
Statistical Analysis 1: Comparison: Group 1 (MPDN+PDN) vs Group 2 (MPDN+PDN+CSA) vs Group 3 (MPDN+PDN+MTX); We used the Kaplan-Meier method to produce survival curves (groups 2 and 3 versus group 1) and compared them with the Log-Rank test. We judged a p value less than 0·05 significant. We reported in the table the incidence rates with 95% confidence intervals of the 3 groups; Test type: Superiority; p = 0.002, Log Rank; Relative risk = 1.65, 95% CI 2-sided [1.24 to 2.14] — RR related to prednisone+methotrexate arm or prednisone+ciclosporin versus prednisone alone
Statistical Analysis 2: Comparison: Group 1 (MPDN+PDN) vs Group 2 (MPDN+PDN+CSA) vs Group 3 (MPDN+PDN+MTX); We used the Kaplan-Meier method to produce survival curves (groups 1 versus groups 2 and 3) and compared them with the Log-Rank test. We judged a p value less than 0·05 significant. We reported in the table the incidence rates with 95% confidence intervals of the 3 groups; Test type: Superiority; p = 0.002, Log Rank; Relative risk = 1.65, 95% CI 2-sided [1.24 to 2.14] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | MPDN+PDN | MPDN+PDN+CSA | MPDN+PDN+MTX
Serious Adverse Events (participants affected / at risk) | 1/47 | 5/46 | 2/46
Other Adverse Events (participants affected / at risk) | 29/47 | 35/46 | 29/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPDN+PDN (N=47) | MPDN+PDN+CSA (N=46) | MPDN+PDN+MTX (N=46)
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermo-hypodermitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MPDN+PDN (N=47) | MPDN+PDN+CSA (N=46) | MPDN+PDN+MTX (N=46)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 8 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 11 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 0
Infection and infestations (Infections and infestations) | 5 | 14 | 14
Cushing syndrome (Endocrine disorders) | 9 | 6 | 9
Weight gain (Metabolism and nutrition disorders) | 3 | 1 | 3
Increases in serum creatinine (Investigations) | 0 | 3 | 3
Headache (Nervous system disorders) | 1 | 5 | 1
General disorders and administration site conditions (Injury, poisoning and procedural complications) | 1 | 9 | 2
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4
Psychiatric disorders (Psychiatric disorders) | 2 | 5 | 4
Metabolic disorders (Metabolism and nutrition disorders) | 3 | 4 | 4
Vascular disorders (Vascular disorders) | 2 | 7 | 1
Tachycardia (Cardiac disorders) | 0 | 3 | 0
Eye disorders (Eye disorders) | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2007-02-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT00323960/Prot_000.pdf